CLINICAL TRIAL: NCT06304792
Title: Immediate Versus Postponed Single Blastocyst Transfer in Programmed or Stimulated Cycle Frozen Embryo Transfer: a Multicenter Randomized Controlled Trial
Brief Title: Immediate Versus Postponed Single Blastocyst Transfer in Programmed or Stimulated Cycle Frozen Embryo Transfer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anja Bisgaard Pinborg, Prof. DMSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-22030591
Record Dates: First submitted 2024-02-23; First posted 2024-03-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Infertility; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate FET in a stimulated or programmed cycle (Experimental): Stimulated or programmed cycle FET is performed in the first cycle following failed fresh embryo transfer or freeze all.
  Interventions: Procedure: Immediate FET in a stimulated or programmed cycle
- Postponed FET in a stimulated or programmed cycle (No Intervention): Stimulated or programmed cycle FET is performed at least one full menstrual, or one hormonal replacement treatment (HRT) cycle in case of oligo-anovulation, after the fresh embryo transfer or freeze-all cycle

INTERVENTIONS:
Procedure: Immediate FET in a stimulated or programmed cycle — Patients will undergo FET in the cycle immediately following oocyte retrieval and a failed fresh embryo transfer or freeze all.
  Arms: Immediate FET in a stimulated or programmed cycle

SUMMARY:
The aim of this randomized controlled trial is to examine whether single blastocyst transfer in the first cycle after oocyte retrieval (immediate) is non-inferior to single blastocyst transfer in a subsequent cycle (postponed) in stimulated or programmed cycle frozen embryo transfer (FET). The primary outcome is live birth rate.

DETAILED DESCRIPTION:
This is a multicenter randomized controlled trial with the aim of investigating if FET in the first cycle after oocyte retrieval (immediate) is non-inferior to the standard treatment where FET is postponed to a subsequent cycle.

Patient inclusion is set to begin in February 2024 and continue til August 2028. A total of 484 patients will be included according to the inclusion and exclusion criteria.

Patients will be randomized 1:1 to either immediate or postponed FET. Randomization is stratified for stimulated FET with letrozole, stimulated FET with gonadotropins and programmed FET (estradiol and progesterone treatment).

The study groups will be:

1. FET immediate: Programmed cycle (PC) or Stimulated cycle (SC) FET in the first cycle after oocyte retrieval and fresh embryo transfer or freeze-all.
2. FET postponed: PC or SC FET after at least one cycle following oocyte retrieval and fresh embryo transfer or freeze-all.

Participants will have a visit on cycle day 2-4 of the first period after oocyte retrieval where baseline characteristics will be assessed. Patients start treatment according to the randomization, thus women in the FET immediate group will start FET immediately whereas women randomized to postponed FET will wait for at least one cycle (natural or induced by sequential estradiol-Provera treatment in oligo-anovulatory women).

SC-FET: Patients undergoing stimulated cycle FET will start the mild ovarian stimulation with either letrozole 5 mg (2,5) daily for five days starting on cd 3-5, or with gonadotropins hMG/rFSH 50-75 IE daily (initial dose may be higher if needed based on previous treatments). Ovulation trigger (hCG) are administered when the leading follicle reaches ≥18 mm (letrozole) or ≥17 mm (gonadotropin). Blastocyst transfer will be performed 6-7 days after trigger.

PC-FET: Patients undergoing PC FET will start treatment with estradiol 6 mg/day from cycle day 3-5, and after 10-12 days an ultrasound scan will be performed. If the endometrial thickness is <7 mm, plasma levels of estradiol can be measured and additional estradiol is added according to local clinical practice. After another 4-6 days a new ultrasound scan is performed and progesterone supplementation will be added no matter of the endometrial thickness and blastocyst transfer will be performed on the 5th or the 6th day of progesterone supplementation.

Blood samples will be drawn on the baseline visit (all patients), on cycle day 2-4 in the postponed FET group, on the day of hCG trigger (SC) or on progesterone supplementation day 10-12 (PC), on the day the blastocyst transfer, and on the day of pregnancy testing.

In case of pregnancy, pregnancy and delivery data will be collected from the patients medical records and the new borns birth record. This will be done in accordance to an informed consent form, which is signed by the participants at inclusion.

The primary outcome of the study will be live birth rates (LBR). Secondary outcomes include 1) LBR per blastocyst transfer 2) Clinical pregnancy rate (CPR) 3) ongoing pregnancy rate (OPR) 4) miscarriage rate (MR) 5) cancelled cycle rate including reason for cycle cancellation 6) endocrinology of the luteal phase by means of hormone levels at predefined time-points 7) number of ovarian follicular structures >10 mm at cycle day 2-5 of the treatment cycle and on the first day of progesterone supplementation 8) time to pregnancy and live birth from start of ovarian stimulation in the fresh cycle.

Pregnancy related complications, such as preeclampsia, pregnancy related hypertension, medically assisted delivery and postpartum hemorrhage (>100 mL), and neonatal outcomes including preterm birth, low birth weight, small or large for gestational age and perinatal mortality, will also be assessed and compared between groups.

An interim analysis will be performed after inclusion of the first 150 patients (n=75 in each group). The mean number of scans will be compared between the two groups. This will be done to evaluate if the mean number of ultrasoundsscans in the intervention group exceeds that of the control group by more than two scans, if this is the case we will consider terminating the trial.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for FET in a programmed- or stimulated cycle immediately following a fresh embryo transfer or freeze all cycle
* Oligo-anovulatory women (cycle length > 35 days)
* Ovulatory women (cycle length 21-35 days)
* At least one vitrified day 5 or 6 blastocyst with Gardner score of ≥ 3BB at the day of vitrification

Exclusion Criteria:

* Uterine malformation
* Presence of hydrosalpinx, submucosal uterine myomas or uterine polyps
* Allergies or contraindication to standard fertility medication
* Male or female HIV or Hepatitis B or C
* Preimplantation genetic testing (PGT) in the fresh cycle
* Testicular sperm aspiration (TESA)
* Severe OHSS with hospital admission and ascites drainage during the fresh cycle
* Oocyte donation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 484 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | One year follow up from positive pregnancy test.
  Live birth rate in immediate FET compared to postponed FET in women undergoing FET in a stimulated or programmed cycle.

SECONDARY OUTCOMES:
Live birth rate per blastocyst transfer | One year follow up from positive pregnancy test.
  Live birth rate overall in both groups
Ongoing pregnancy rate | At 7 or 8 weeks of gestation in case of pregnancy
  Ongoing pregnancy rate where pregnancy is assessed by ultrasound in the immediate versus the postponed group
Miscarriage rate | Until 22 weeks of gestation in women with positive pregnancy test
  Rate of pregnancy loss in the immediate versus the postponed group
Cancelled cycle rate and reason for cancelled cycles | Will be assessed through study participation dependent on the participants cycle up to 50 days
  Cancelled cycle rate in the immediate versus the postponed group
Endocrinology of the luteal phase | Through each participants cycle, will be dependent on participants cycle up to 50 days
  Hormone levels at predefined time-points in the immediate versus the postponed group
Number of ovarian follicular structures >10 mm | Twice through the cycle, dependent on participants cycle length up to 50 days
  Number of ovarian follicular structures >10 mm in the immediate versus postponed arm
Time-to-pregnancy | From day of ovarian stimulation until clinical pregnancy dependent on participants cycle length up to 70 days
  Time-to-pregnancy in the immediate versus postponed arm
Time-to-live-birth | From day of ovarian stimulation through study completion up to 1 year
  Time-to-live-birth in the immediate versus postponed arm
Pregnancy related complications | One year follow up from positive pregnancy test
  Pregnancy related complications in patients receiving immediate versus postponed FET
Neonatal outcomes (weight in kilograms) | One year follow up from positive pregnancy test
  Neonatal outcome in children of patients in patients receiving immediate versus postponed FET
Neonatal outcomes (length in cm) | One year follow up from positive pregnancy test
  Neonatal outcome in children of patients in patients receiving immediate versus postponed FET
Neonatal outcomes (apgar score at 1, 5 and 10 minutes postpartum) | One year follow up from positive pregnancy test
  Neonatal outcome in children of patients in patients receiving immediate versus postponed FET. The apgar score is reported on a scale of 0-10, 10 being the highest score.
Quality of life based on the Copenhagen Multicenter Psychosocial Infertility (COMPI) stress scale questionnaires | Questionnaires will be handed out at baseline and after blastocyst transfer timeframe will depend on the participants cycle up to 50 days
  Quality of life in the immediate versus postponed arm. Reported on scales of "excellent, very good, good, fair or poor" or on a scale of "all the time, most of the time, sometimes, a little of the time, none of the time".

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Departmen, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
In case of requests, the final data will be shared according to the ICJME guidelines. Sharing will only be done with parties presenting new research projects which have been approved by the steering committee of the research team. Any new project involving data collected in this trial must also be approved by Danish authorities. Expenses for data sharing will be covered by those requesting it. Data will not be shared with research groups conducting projects with the same aim, secondary aims and/or purposes as ours until three months after publication of the primary and secondary outcomes of this study.
Supporting Information: Study Protocol
Time Frame: From 3 months after publication on the primary and secondary outcomes in this study.

REFERENCES:
- [Derived] Colombo C, Johansen AS, Saupstad M, Bergenheim SJ, Dam TV, Wang NF, Oxlund-Mariegaard B, Lokkegaard E, Husth M, Lauritsen MP, Forman JL, Freiesleben NC, Nohr B, Lossl K, Pinborg A. Immediate versus postponed blastocyst transfer in stimulated or programmed frozen embryo transfer cycles - a protocol for a non-blinded randomised clinical trial. Dan Med J. 2025 Jul 22;72(8):A03250214. doi: 10.61409/A03250214. PMID 40747727